CLINICAL TRIAL: NCT00355420
Title: Evaluation of the Change in Length of the Femur and Tibia in Children After Treatment of Femur Fractures With External Fixators, Plaster of Paris or Internal Fixation
Brief Title: Evaluation of the Change in Length of the Leg in Children After Treatment of Femur Fractures.
Status: Withdrawn | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: LLD01-HMO-CTIL
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Fractures
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Femur fractures are a common injury in the Pediatric population. Despite their high incidence little do we know about the long term implications on the bones' length. Our main goal is to clarify this obscure issue by assessing the femoral and tibial length as determined by the fractures, measuring techniques and treatment modalities

ELIGIBILITY:
Inclusion Criteria:

* Males between the ages 0-16.
* Females between the ages 0-14.
* Signed Informed consent

Exclusion Criteria:

* A refusal by the patient or his legal guardian to continue the follow-up with the
* Pediatric Orthopedic clinic, or to have the CT scanograms.
* Patients with severe contractures in the lower extremities
* Patients with multiple lower extremity fractures
* Pregnancy

Max Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children that sufferinf from LLD
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Ron Lamdan, Dr., Principal Investigator — Hadassah Medical Organization; Shlomo Porat, Prof., Study Chair — Hadassah Medical Organization; Naum Simanovski, Dr., Study Director — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel